CLINICAL TRIAL: NCT02925455
Title: Contralaterally Controlled Functional Electrical Stimulation for Hand Opening in Hemiplegic Cerebral Palsy: Pilot Randomized Controlled Trial
Brief Title: Contralaterally Controlled FES for Hand Opening in Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: The Cleveland Clinic (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michael Fu, Assistant Professor, Physical Medicine and Rehabilitation, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-400; 1R21HD088987-01 (NIH)
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Cerebral Palsy
Keywords: Hemiplegia; Functional Electrical Stimulation; Video Games; Occupational Therapy
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulation + Video Games (Experimental): Contralaterally-controlled functional electrical stimulation (CCFES) enables patients with upper extremity hemiplegia to open their paretic hand by stimulating finger and thumb extensors with surface electrodes. CCFES is used during functional task practice and hand therapy video games to link motor intent with execution. Four intuitive and engaging games were developed to provide goal-oriented motor skill training, impairment-appropriate difficulty, and performance feedback that motivates iterative play and skill improvement.
  Interventions: Device: Contralaterally-controlled functional electrical stimulation; Device: Hand therapy video games
- Video Games (no stimulation) (Active Comparator): Participants receive duration-matched, identical hand therapy video games and task practice therapy as the experiment arm, but do not receive CCFES to assist hand opening.
  Interventions: Device: Hand therapy video games

INTERVENTIONS:
Device: Contralaterally-controlled functional electrical stimulation — Contralaterally-controlled functional electrical stimulation (CCFES) is electrical stimulation of weak muscles of an impaired limb controlled via movement of the unimpaired contralateral limb.
  Arms: Stimulation + Video Games
Device: Hand therapy video games — Hand therapy video games are designed to provide therapy to weak muscles of an impaired limb via goal-directed movements.

SUMMARY:
This is a pilot randomized controlled trial of an intervention to improve arm function in children ages 6 to 17 with cerebral palsy and upper limb hemiparesis. Twenty participants will be randomized to either a group treated with neuromuscular electrical stimulation and video games or video games alone. Both groups will receive 6 wks of treatment consisting of home and lab sessions. Both the experiment group and control group interventions consist of therapist-guided sessions in the rehabilitation clinic and self-administered or caregiver-assisted sessions at home. While both groups will receive the same task practice and video game training, only the experiment group will receive an electrical stimulation device to assist with hand opening during practice. Changes in upper extremity motor impairment and function will be assessed for each participant at baseline, mid treatment, end of treatment and at 3 mo follow-up.

DETAILED DESCRIPTION:
Rehabilitation clinic sessions - These will occur up to twice per week for the first 3 weeks and once per week for the second 3 weeks of the 6 week treatment. They are therapist-guided and last up to 90 min consisting of 45 minutes of contralaterally-controlled functional electrical stimulation (CCFES)-mediated video games and up to 45 minutes of CCFES-mediated functional task practice. Early sessions will focus on training the patient and caregiver to self-administer play of a CCFES-mediated video game at home. As proficiency with one game develops, more games will be introduced. The functional task practice part of the session will engage the participant in using the CCFES system to assist them in practicing using their hand in activities such as lacing beads, throwing balls, eating finger foods, and other play and activities of daily living. Prior to the start of lab treatment, the investigators will assess hand extensor and flexor muscle co-activation (see below).

Home sessions - These consist of CCFES-mediated hand opening and video game exercises with caregiver assistance and supervision as needed. As proficiency develops and more games are added, each home session will increase in duration up to 90 minutes per day, as determined by the treating therapist based on the adherence of each participant. Self report of game difficulty and engagement will be made at the completion of each game (see below)

ELIGIBILITY:
Inclusion Criteria:

* Upper Extremity hemiparesis from Cerebral Palsy
* Age 6-17
* Caregiver can transport participant to weekly sessions and assist with home treatment
* Medically stable; stable medications
* Recall 2 of 3 items after 30 min
* Finger extension strength ≤ 4/5 on paretic side
* Able to follow 3-stage commands
* Adequate active movement of paretic arm to position the hand for table-top task practice
* Skin intact on hemiparetic arm
* Surface neuromuscular electrical stimulation trial opens hand without pain
* Full volitional hand opening and closing of contralateral hand
* Box & Blocks Score of weaker side < 90% of stronger side score
* Able to hear and respond to auditory cues
* English proficiency of both caregiver and child

Exclusion Criteria:

* Uncontrolled seizure disorder
* Co-existing neurological conditions other than cerebral palsy affecting the hemiparetic upper limb (e.g., peripheral nerve injury, Parkinson's disease, spinal cord injury, traumatic brain injury, multiple sclerosis, stroke, hemispherectomy)
* Severely impaired cognition and communication
* History of cardiac arrhythmias with hemodynamic instability
* Insensate arm, forearm, or hand
* Uncompensated hemi-neglect
* Cardiac pacemaker or any other implanted electronic systems
* Pregnant
* Intramuscular Botox injections in any upper extremity muscle in the last 3 months
* Severe visual impairment

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2016-10-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Fu, PhD, Principal Investigator — MetroHealth Medical Center
Locations (2):
- United States (2):
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stimulation + Video Games | Video Games (no Stimulation)
Started | 9 | 6
Completed | 7 | 6
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stimulation + Video Games | Video Games (no Stimulation) | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.22 (2.86) | 12.17 (4.31) | 11.60 (3.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 7 | 4 | 11
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Manual Ability Classification System [Count of Participants; unit: Participants]
  Level I: Level 1: Objects are handled easily and successfully | 0 | 0 | 0
  Level 2: Handles most objects but with some reduced quality and/or speed | 6 | 4 | 10
  Level 3: Handles objects with difficulty - child will need help to prepare and/or modify activities | 3 | 2 | 5
  Level 4: Handles limited selection of easily managed objects and always requires some help | 0 | 0 | 0
  The child is not able to handle objects or to complete even simple actions with their hands | 0 | 0 | 0
Delivery Type [Count of Participants; unit: Participants]
  Vaginal | 4 | 2 | 6
  Cesarean | 5 | 4 | 9
Affected Hand [Count of Participants; unit: Participants]
  Right | 5 | 4 | 9
  Left | 4 | 2 | 6
Time of injury [Count of Participants; unit: Participants]
  Perinatal | 2 | 0 | 2
  Postnatal | 1 | 1 | 2
  Prenatal | 4 | 3 | 7
  Unknown | 2 | 2 | 4
Presence of Prenatal Complications [Count of Participants; unit: Participants]
  Yes | 2 | 2 | 4
  No | 7 | 4 | 11
Lesion Type [Count of Participants; unit: Participants]
  Cystic Encephalomalacia | 1 | 0 | 1
  Encephalomalacia | 1 | 1 | 2
  Hemorrhagic | 3 | 2 | 5
  Ischemic | 1 | 0 | 1
  Periventricular Leukomalacia | 1 | 0 | 1
  Unknown | 2 | 3 | 5
Lesioned hemisphere [Count of Participants; unit: Participants]
  Bilateral | 2 | 0 | 2
  Left | 4 | 3 | 7
  Right | 2 | 2 | 4
  Unknown | 1 | 1 | 2
Hand Dominance [Count of Participants; unit: Participants]
  Right | 4 | 3 | 7
  Left | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Assisting Hands Assessment Logit Score at End of Treatment
Description: Participants played a game that required them to perform bimanual tasks while being video recorded. The amount of involvement of the affected arm is scored by viewing the video and converted into a logit score (0-100), with a higher value indicating a better outcome.
Time Frame: 2 time points: prior to treatment and at end of 6 weeks of treatment
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Stimulation + Video Games | Video Games (no Stimulation)
Number analyzed (Participants) | 9 | 6
Scores on a scale | 2.63 [0.415 to 4.85] | 4.33 [2.44 to 6.23]

2. Secondary Outcome: Change in Melbourne 2 Motor Assessment at End of Treatment
Description: Participants perform 14 test tasks that require reach, grasp, release, and manipulation of simple objects. A video of the test is recorded for scoring across the 30 score items using a three, four or five point scale (higher values indicating better outcomes). Item scores relating to four elements of movement are measured and summed within the corresponding sub-scale. A percentage of the total score (range 0-100%) for each subscale is computed and reported separately, with higher values indicating better outcomes.
Time Frame: 2 time points: prior to treatment and at end of 6 weeks of treatment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Stimulation + Video Games | Video Games (no Stimulation)
Number analyzed (Participants) | 9 | 6
units on a scale
  Range of Movement (higher values indicate greater shoulder, trunk, elbow, forearm range of motion) | 3.50 [-2.20 to 9.19] | 6.17 [0.106 to 12.2]
  Target Accuracy (higher values indicate closer initial point of sustained contact with objects) | 1.91 [-4.63 to 8.45] | -2.00 [-10.1 to 6.08]
  Dexterity (higher values indicate greater grasp, release, and manipulation ability) | 9.49 [0.317 to 18.7] | 7.02 [-0.413 to 14.5]
  Fluency (higher values indicate smother, more coordinated motion) | 6.39 [-2.99 to 15.8] | 3.97 [-0.253 to 8.19]

3. Other Pre Specified Outcome: Change in Box and Block Test Score at Treatment End
Description: The Box and Blocks test counts how many times the participant can pick up 1 block at t time, move it over a partition, and release it in a target area within 60 seconds.
  The minimum score is 0. There is no maximum score. The average score of healthy individuals within the age range of this study ranges from 70 to 79.
  Higher scores are considered to be a better outcome. For each individual, the score prior to treatment was subtracted from the score at 6 months after completion of treatment. Then for each treatment group, these change scores were averaged.
Time Frame: 2 time points: prior to treatment and after 6 weeks of treatment
Measure: Mean (95% Confidence Interval); unit: Number of blocks
Arm/Group | Stimulation + Video Games | Video Games (no Stimulation)
Number analyzed (Participants) | 9 | 6
Number of blocks | 2.47 [-1.88 to 6.81] | 0.667 [-1.85 to 3.19]

4. Other Pre Specified Outcome: Change in Instrumented Sine Wave Finger Tracking Error at Treatment End
Description: Finger movement tracking is a method of measuring motor control. The degree of finger extension will be displayed as a cursor on a computer screen, its vertical position corresponding to the degree of finger extension. A sinusoidal trace having a frequency of 0.1 Hz (1 cycle in 10 seconds) will scroll across the screen. The amplitude of the sine-wave track will be scaled so that it oscillates between 15% and 85% of the participant's full active finger extension. The participant will be seated with the wrist and forearm stabilized in a neutral posture. The participant's task is to keep the cursor on or as close to the scrolling trace as possible by extending and flexing their index finger. The vertical distance between the cursor and the target trace will be calculated for every time point of data collected. The error for each 30-sec trial will be the average vertical distance that is equivalent to a percentage of volitional range of motion.
Time Frame: 2 time points: prior to treatment start and at end of treatment week 6.
Measure: Mean (95% Confidence Interval); unit: Percentage of range of motion
Arm/Group | Stimulation + Video Games | Video Games (no Stimulation)
Number analyzed (Participants) | 9 | 6
Percentage of range of motion | -3.59 [-5.51 to 01.67] | -3.36 [-6.21 to -0.510]

5. Other Pre Specified Outcome: Number of Cumulative Hand Movement Repetitions During Game Play
Description: The number of hand movement repetitions was computed by calculating the number of hand trajectory direction changes divided by two.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Number of hand movement repetitions
Arm/Group | Stimulation + Video Games | Video Games (no Stimulation)
Number analyzed (Participants) | 7 | 6
Number of hand movement repetitions | 22095 (7385.2) | 23035 (16169)

ADVERSE EVENTS:
Time Frame: Up to 18 weeks (from baseline to 12 weeks after end of the 6-week treatment)
Arm/Group | Stimulation + Video Games | Video Games (no Stimulation)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT02925455/Prot_SAP_000.pdf